CLINICAL TRIAL: NCT03082846
Title: Treatment of High-grade Gliomas Using Escalating Doses of Hypofractionated Simultaneous Integrated Boost-intensity Modulated Radiation Therapy in Combination With Temozolomide - a Modified Phase I Clinical Trial
Brief Title: Treatment of High-grade Gliomas Using Hypofractionated Radiation Therapy -a Phase I Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xue Xiaoying (Other)
Responsible Party: Sponsor-Investigator, Xue Xiaoying, Department of Radiotherapy, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: phase I clinical trial-gliomas
Record Dates: First submitted 2017-02-22; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Glioma; Radiotherapy, Intensity-Modulated; Maximum Tolerated Dose
Keywords: malignant glioma; intensity modulated radiation therapy; simultaneous integrated boost; hypofractionation; temozolomide; maximum tolerated dose
MeSH Terms: conditions — Glioma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypofractionated group (Experimental): hypofractionated group using hypofractionated radiation with temozolomide chemotherapy: Malignant gliomas patients received concurrent postoperative radiotherapy and chemotherapy.Intensity-modulated radiotherapy is adopted, the dose at each fraction is gradually increased from 2.8 Gy/f (total of 20 times) with an escalating dose interval of 0.4 Gy in PTV1. The planning target volume (PTV2) remain unchanged with 2.5 Gy each time and a total of 50 Gy/20 f. Temozolomide is administered orally every day at 75 mg/m2 during radiotherapy and at 150-200 mg/m2 for 12 cycles following completion of chemoradiotherapy.
  Interventions: Radiation: hypofractionated radiation; Drug: Temozolomide chemotherapy

INTERVENTIONS:
Radiation: hypofractionated radiation — The simultaneous integrated boost-intensity modulated technology is adopted to increase both the dose in the surgical cavity and residual tumor (PTV1).The dose at each fraction is gradually increased from 2.8 Gy/f (total of 20 times) with an escalating dose interval of 0.4 Gy in PTV1, until dose-limiting toxicity is present,the highest target single dose is 4 Gy/f. The planning target volume (PTV2) including the 2 cm region around surgical cavity and residual tumor remain unchanged, with 2.5 Gy each time and a total of 50 Gy/20f.
Drug: Temozolomide chemotherapy — Temozolomide(TMZ) is administered orally every day at 75 mg/m2 during radiotherapy and at 150-200 mg/m2 for 12 cycles following completion of chemoradiotherapy.
  Other Names: TMZ chemotherapy

SUMMARY:
Postoperative conventional radiation at 60 Gy/30f is currently still considered the standard radiotherapy mode for high-grade gliomas; however, the efficacy is still unsatisfactory. Studies in recent years have shown that hypofractionated simultaneous integrated boost-intensity modulated radiation therapy (SIB-IMRT) has certain survival benefits over other fractionation methods; but, the best hypofractionation mode and its efficacy have not been confirmed. The purpose of this study is to investigate the maximum tolerated dose (MTD) of hypofractionated SIB-IMRT with stepwise escalating of doses combined with temozolomide (TMZ) for the treatment of malignant gliomas.

DETAILED DESCRIPTION:
Background: Postoperative conventional radiation at 60 Gy/30f is currently still considered the standard radiotherapy mode for high-grade gliomas; however, the efficacy is still unsatisfactory. Studies in recent years have shown that hypofractionated simultaneous integrated boost-intensity modulated radiation therapy (SIB-IMRT) has certain survival benefits over other fractionation methods; but, the best hypofractionation mode and its efficacy have not been confirmed. The purpose of this study is to investigate the maximum tolerated dose (MTD) of hypofractionated SIB-IMRT with stepwise escalating of doses combined with temozolomide (TMZ) for the treatment of malignant gliomas. Methods: Malignant gliomas patients receive concurrent postoperative radiotherapy and chemotherapy. The simultaneous integrated boost-intensity modulated technology is adopted to increase both the dose in the surgical cavity and residual tumor (PTV1). The dose at each fraction is gradually increased from 2.8 Gy/f (total of 20 times) with an escalating dose interval of 0.4 Gy. The planning target volume (PTV2) including the 2cm region around surgical cavity and residual tumor remain unchanged, with 2.5 Gy each time and a total of 50 Gy/20f. The subsequent group of patients is advanced to the next dose level until dose-limiting toxicity (DLT) is present. The dose, one level lower than the DLT, is the MTD. The highest target single dose is 4 Gy/f. TMZ is administered orally every day at 75 mg/m2 during radiotherapy and at 150-200 mg/m2 for 12 cycles following completion of chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative grades III and IV glioma patients confirmed by pathology.
2. The ages are between 18-70 years.
3. Karnofsky performance score（KSP）≧60.
4. Expected survival period ≧3 months.
5. Blood routine and liver and kidney functions are normal.
6. Receive cranial MRI examination after 48 h of surgery.
7. Radiotherapy is performed after 2-4 weeks of surgery.
8. Patients with restricted lesions and non-diffuse growth.
9. Maximum diameter of the residual tumor, surgical cavity, and primary tumor bed are ≦6 cm.

Exclusion Criteria:

1. Lesions are in the brain stem and thalamus.
2. Pregnant and lactating women.
3. Secondary primary malignant tumor.
4. Severe pulmonary infection.
5. Combination with mental illness or another disease that require hospitalization.
6. Patients had received chemotherapy or brain radiotherapy previously.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2016-12-03 (Actual)

PRIMARY OUTCOMES:
the maximum tolerated dose(MTD) | 1year
  Safety and tolerability of hypofractionated simultaneous integrated boost intensity modulated radiation therapy (SIB-IMRT) combined with standard temozolomide chemotherapy.
  The maximum tolerated dose of hypofractionated radiation combined with concurrent temozolomide in newly diagnosed highgrade glioma is being explored.

SECONDARY OUTCOMES:
Progression free survival | 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoying xue, doctor, Study Director — Department of Radiotherapy

IPD SHARING:
Plan to Share IPD: No